CLINICAL TRIAL: NCT00257738
Title: A Phase 1 Open Label, Dose Escalation Study to Evaluate the Effect of Four Doses of MAGE-A3/HPV 16 Trojan Peptides 0001 and 0002 Administered Subcutaneously in Combination With Montanide and GM-CSF on Immunological Response, Safety, Tolerability, and Preliminary Efficacy in Patients With Squamous Cell Carcinoma of the Head and Neck
Brief Title: 0804 GCC: MAGE-A3/HPV 16 Vaccine for Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00041372; R01DE015324 (NIH); NCT00704041 (obsolete NCT alias)
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — MAGEA3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAGE -A3 vaccine (Experimental): for those individuals in which tumor tests positive for MAGE-A3
  Interventions: Biological: MAGE-A3
- HPV 16 vaccine (Experimental): for patients with HPV 16 positive tumor
  Interventions: Biological: HPV-16 vaccine

INTERVENTIONS:
Biological: MAGE-A3 — Three dose levels of MAGE-A3 vaccine will be tested : 500ug, 1000 ug and 1500 ug
  Arms: MAGE -A3 vaccine
Biological: HPV-16 vaccine — Three dose levels of HPV- 16 vaccine will be tested : 500ug, 1000 ug and 1500 ug
  Arms: HPV 16 vaccine

SUMMARY:
Squamous Cell Carcinoma of the Head and Neck (SCCHN) is a devastating illness, the treatment of which is associated with significant morbidity. This type of cancer affects 43,000 individuals each year with an estimated survival rate of 50%. A potential treatment alternative for this patient population is the use of peptide-based immunotherapy. This clinical tial will be using a vaccines comprised on the Trojan peptides MAGE-A3 and HPV 16 to treat patients with Squamous Cell Carcinoma of the Head and Neck who have recurrent, progressive or metastatic SCCHN.

DETAILED DESCRIPTION:
Squamous Cell Carcinoma of the Head and Neck affects 43,000 individuals in the United States annually with an estimated overall survival rate of 50%. In order to improve both the survival rate and quality of life for patients who develop unresectable disease recurrence, new therapeutic alternatives are mandated. One potential treatment alternative for this patient population is the use of peptide-based immunotherapy. Despite the success fo preclinical studies using peptide vaccines, therapeutic responses in patients have been sporadic. The reasons for failure are multifactorial and include problems with patient selection, a limited number of antigenic targets, and an inability to correlate immunologic response with therapeutic efficacy. Specifically, patients with disseminated SCCHN have defects in antigen processing, presentation and effector mechanisms that limit their ability to respond to T cell based immunotherapy. Additionally, a paucity of antigenic peptide epitopes are defined for SCCHN, and immunologic monitoring does not correlate well with clinical response.

Recently several investigators, including our research team, have identified a high prevalence of MAGE-A3 and HPV 16 on SCCHN, and characterized several putative cytolytic and helper epitopes. Additionally, we have defined a novel method to enhance the immune response to therapeutic peptide vaccines using Trojan complexes composed of CD4 and CD8 T-cell epitopes, connected by furin cleavable linkers.

In order to define the feasibility and safety of these agents in combination with GM-CSF and montanide ISA 51 for the immunotherapy of SCCHN, in this proposed trial, we will screen patients for immunologic competence based on specific eligibility criteria including both antigen and HLA-A2 expression on tumors. In registered patients, we will test the ability of two novel Trojan peptide complexes, composed of MAGE-A3 and human papilloma virus 16 (HPV 16) epitopes, to stimulate antigen-specific CD 4 and CD 8 T-cell responses. Finally, we will correlate immunologic response with cell dose and the generation of both HPV 16 and MAGE-A3 antigen loss and HLA-A2 loss variants on tumors by evaluating patients for: 1) Changes in tumor size by both physical measurement and CT plus PET measurement; 2) Determining what proportions of individuals who achieve a complete response (CR), partial response (PR), or have stable disease (SD); 3) Progression-free survival; 4) Survival. Successful completion of this clinical trial will result in the development of a strong foundation for a Phase II/III clinical trial using HPV 16 and MAGE-A3 Trojan peptides for the immunotherapy of SCCHN.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Biopsy proven progressive, recurrent (post-surgical, radiation therapy, chemotherapy, combination therapy),or metastatic SCC of the head and neck which, in the judgment of the attending physician, is incurable by standard treatment modalities, OR Biopsy proven SCC which the patient is unwilling to have treated with surgery, chemotherapy or radiation therapy
3. One or more of the following: -MAGE-A3 positive tumor -HPV 16 positive tumor.
4. Laboratory values obtained less than or equal to 30days prior to registration: -Alkaline phosphatase less than or equal to 3x upper normal limit (UNL) -AST less than or equal to 3x UNL -Creatinine less than or equal to 1.5 x UNL -Hemoglobin greater than or equal to 9.0 g/dL -Albumin greater than or equal to 3 mg/dL
5. The subject must be capable of understanding the investigational nature, potential risks and benefits of the study and capable of providing valid informed consent.
6. The subject must be willing to return to the University of Maryland Medical center for treatment and study related follow up procedures including blood and tumor collections and completion of imaging studies as required by the protocol.
7. ECOG performance status 0-2.
8. Tumor that is biopsy accessible and measurable. This includes, but is not limited to, open biopsy, endoscopic biopsy, image guided biopsy, core biopsy and fine needle aspiration.

EXCLUSION

1. Any of the following:

   a. Known HIV infection, b. Other circumstances (i.e. concurrent use of systemic immunosuppressants and immunocompromising condition) that in the opinion of the physician renders the patient a poor candidate for this trial. c. Patients with ANY malignant or metastatic SCC mass or lesion within the Central Nervous System (CNS). (e.g. Intraparenchymal/ Brain, Intracordal / Spinal Canal, Bony masses or lesions with extension into the CNS parenchyma) d. Patients with ANY malignant or metastatic SCC mass or lesion or a volume of a mass or lesion in a location that in the judgment of the investigator may significantly impair the health of or threaten the patients life, should an Inflammatory Response occur.
2. Any of the following prior therapies: Chemotherapy less than or equal to 4 weeks prior to registration Immunotherapy less than or equal to 4 weeks prior to registration Biologic therapy less than or equal to 4 weeks prior to registration Radiation therapy less than or equal to 4 weeks prior to registration
3. Any of the following: Pregnant women Nursing women unwilling to stop breastfeeding Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.) NOTE:This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.
4. Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation).
5. Either of the following: Other active cancer requiring therapy to control the disease History of other malignancy (i.e. excluding disease under study) within 3 years Exceptions to the above include: adequately treated basal cell or squamous cell skin cancer, prostate cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing toxicity | 2 year
  Maximum grade of each toxicity and percentage of patients experiencing toxicity as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Tumor response | 4 years
  Tumor response as assessed by RECIST
Tumor infiltrating lymphocytes | 4 years
  analysis will be performed to assess the degree of tumor infiltration by lymphocytes per- and post treatment (if possible)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Edelman, MD, Principal Investigator — University of Maryland, Greenebaum Cancer Ctr
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States